CLINICAL TRIAL: NCT02068482
Title: Evaluation of Immunohistological Pattern in Patients With Uncomplicated Symptomatic Diverticular Disease and Correlation Between Intraluminal Bacterial Flora and Phlogosis
Brief Title: Immunohistology in USDD and Correlation Between Bacterial Flora and Phlogosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Director of Digestive and Surgical Endoscopy, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDSNC2009
Record Dates: First submitted 2014-02-12; First posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Diverticular Disease
Keywords: Uncomplicated; Symptomatic
MeSH Terms: conditions — Diverticular Diseases | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1a USDD (Active Comparator): Rifaximin 200 mg 6 tbs per day per 15 days/ month for 2 months
  Interventions: Drug: Rifaximin
- 1b USDD (No Intervention): Patients control, no drug
- Control group (No Intervention): Control Group, no disease, no drug

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 200 mg 6 tbs per day per 15 days/ month for 2 months
  Other Names: Normix
  Arms: 1a USDD

SUMMARY:
Diverticulosis of the colon is a frequent condition in adults in western countries and a significant number of patients experience clinical symptoms even when the diverticulosis is not complicated by diverticulitis.

Both central and mucosal immunity are altered in Uncomplicated Symptomatic Diverticular Disease (USDD) and Rifaximin ameliorate clinical symptoms and normalize the immunological abnormalities.

The Study Protocol is verify the modifications in the immunological pattern induced by reducing bacteria related activation of immunity by Rifaximin treatment.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age 18 or more
* radiologic or endoscopic diagnosis of diverticular disease located in sigma or colon descendent
* Informed consent
* patients willing to participate in to the study

Exclusion Criteria:

* other colon diseases
* Inflammatory Bowel Diseases
* signs or symptoms of inflammation
* consumption of : antibiotics, anti-inflammatory drugs ( FANS and 5-ASA), prebiotics, Proton Pump Inhibitors, corticosteroids, fiber within three months
* pregnancy and breast feeding
* acute diverticulitis characterized by:
* moderate/sever pain in left iliac fossa
* fever > 38°C
* abdominal pain
* haematochezia
* leukocytosis (20% more than the normal range)
* remote acute diverticulitis
* rifaximin hypersensitivity
* neoplastic diseases
* immunodeficiencies
* poor physical conditions
* leaver deficiencies (Child C), kidney (Creatinine>2,2 mg/dl), heart (NYHA 3-4)
* major psychiatric illness
* drugs abuses and alcoholism
* participations in other clinical trials within 4 weeks
* patients unwillingness certificate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Immunohistological Pattern | Two months
  Lymphocytes in peripheral Blood, Lymphocytes in the Sigmoid Mucosa, Lymphocytes in the Transverse Mucosa, Monocytes and Granulocytes in Peripheral Blood

SECONDARY OUTCOMES:
Clinical Symptoms | Two Months
  Dyspepsia, Meteorism, Abdominal pain, Tenesmus, Diarrhea, Fever, Fever with Chills, Painful Palpation, VAS, Likert, Numbers of Evacuations

CONTACTS AND LOCATIONS:
Overall Officials: Franco Pandolfi, Professor, Principal Investigator — CU Sacred Heart; Lucio Petruzziello, Doctor, Study Chair — CU Sacred Heart; Paola Cesaro, Doctor, Study Chair — CU Sacred Heart; Rossella Cianci, Doctor, Study Chair — CU Sacred Heart
Locations (1):
- Cattholic University of the Sacre Heart, Rome, Italy, Italy

REFERENCES:
- [Derived] Cianci R, Frosali S, Pagliari D, Cesaro P, Petruzziello L, Casciano F, Landolfi R, Costamagna G, Pandolfi F. Uncomplicated diverticular disease: innate and adaptive immunity in human gut mucosa before and after rifaximin. J Immunol Res. 2014;2014:696812. doi: 10.1155/2014/696812. Epub 2014 Jul 16. PMID 25133198